CLINICAL TRIAL: NCT04010019
Title: The Impact of Facebook Support Groups for Adults With Chronic Pain: A Randomized Clinical Trial
Brief Title: The Facing Pain Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Mark A. Lumley, Distinguished Professor and Director of Clinical Psychology Training, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 012119B3E
Record Dates: First submitted 2019-06-12; First posted 2019-07-08 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Interested adults will be screened, and eligible participants will be randomly assigned to one of two conditions: a Facebook group for individuals in pain similar to the groups that are occurring naturally (control condition) or an enhanced Facebook group for individuals in pain that is moderated by clinicians and offers psychosocial pain intervention techniques (experimental condition).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Facebook Condition (Experimental): The enhanced Facebook group will be moderated by clinicians and offer psychosocial pain management techniques.
  Interventions: Behavioral: Enhanced Facebook Condition
- Control Facebook Condition (Active Comparator): In the control condition, there will be no outside intervention; rather, the investigators will instruct participants to offer mutual support for the duration of the group and will not comment further.
  Interventions: Behavioral: Control Facebook Condition

INTERVENTIONS:
Behavioral: Enhanced Facebook Condition — The intervention (enhanced Facebook condition) will consist of several training components that were selected based on pain research and platform affordances. The first component will be psychoeducation on pain neurobiology. Emotional validation training will follow. The third component will consist of facilitating patients' emotional disclosure about their pain journeys and lives. The fourth and final intervention component will include prompts to engage participants in activities that they have been avoiding because of their pain.
  Arms: Enhanced Facebook Condition
Behavioral: Control Facebook Condition — The control condition will instruct participants to offer mutual support and will not offer psychosocial intervention.
  Arms: Control Facebook Condition

SUMMARY:
This randomized trial will create and compare two private Facebook conditions for patients with chronic pain. The control condition will be comprised of groups of patients who communicate without much clinician / moderator input, and the experimental condition will have a clinician moderating and teaching patients several techniques designed to facilitate social disclosure, validation, and emotional engagement with avoided activities.

DETAILED DESCRIPTION:
This study will investigate the effectiveness of a private Facebook group for individuals in chronic pain. Currently, more than 100,000 individuals with chronic pain (ICPs) participate in Facebook groups, seeking support from others in similar situations. There are currently some online self-management programs for ICPs; however, most lack a peer support aspect, as they are individualized, self-directed, and focus on instructing patients in how to manage their pain. The goals of the proposed online pain support group are: 1) to provide peer-to-peer social support for individuals with chronic pain; and 2) to disseminate psychosocial pain management techniques using a social media platform. Screened participants will be assigned to one of two conditions: a Facebook group similar to the groups that are occurring naturally (control condition) or an enhanced Facebook group that is moderated by clinicians and offers psychosocial pain management techniques (experimental condition). Both conditions involve peer-to-peer healthcare and support, but the experimental group additionally includes components such as psychoeducation about pain neuroscience, emotional validation training, guided emotional disclosure, and activities to overcome emotional and behavioral avoidance. Findings from this study will offer important information about the impact of Facebook support groups on pain outcomes, and test whether psychosocial pain interventions can be disseminated using a social media platform.

ELIGIBILITY:
Inclusion Criteria:

* Must have chronic pain (i.e., pain that persists for greater than 3 months)
* Must be fluent at reading and writing in English
* Must have an active Facebook account and check Facebook at least 3 times a week

Exclusion Criteria:

* Terminal illness such as cancer
* Active psychosis (e.g., hallucinations, delusions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2020-04-13 (Actual)

PRIMARY OUTCOMES:
Change in pain severity from baseline to post-intervention to 1-month follow-up: Brief Pain Inventory | Pain severity will be assessed at 3 timepoints: 1) baseline (i.e., at the start of the intervention), 2. post-intervention (i.e., immediately after the intervention), and 3. 1-month follow-up (30 days after the intervention ends)
  Brief Pain Inventory (Cleeland, 1991): Pain severity items: 1) Worst pain (0 [no pain] - 10 [pain as bad as you can imagine]), 2) Average pain (0 [no pain] - 10 [pain as bad as you can imagine]), 3) A composite of the 4 pain items (a mean pain severity score) will also be computed (0 [no pain] - 10 [pain as bad as you can imagine])
Change in pain interference from baseline to post-intervention to 1-month follow-up: Brief Pain Inventory | Pain interference will be assessed at 3 timepoints: 1) baseline (i.e., at the start of the intervention), 2. post-intervention (i.e., immediately after the intervention), and 3. 1-month follow-up (30 days after the intervention ends)
  Brief Pain Inventory (Cleeland, 1991): Pain interference items: A composite of the 7 interference items (a mean interference score) will be computed (0 [does not interfere] - 10 [completely interferes])

SECONDARY OUTCOMES:
Change in depression from baseline to post-intervention to 1-month follow-up | Depression will be assessed at 3 timepoints: 1) baseline (i.e., at the start of the intervention), 2. post-intervention (i.e., immediately after the intervention), and 3. 1-month follow-up (30 days after the intervention ends)
  PROMIS Emotional Distress - Depression - Short Form 8a v1.0: A composite of the 8 depression items (a mean depression score) will be computed (1 [low depression score] - 5 [high depression score])
Change in anxiety from baseline to post-intervention to 1-month follow-up | Anxiety will be assessed at 3 timepoints: 1) baseline (i.e., at the start of the intervention), 2. post-intervention (i.e., immediately after the intervention), and 3. 1-month follow-up (30 days after the intervention ends)
  PROMIS Emotional Distress - Anxiety - Short Form 8a v1.0: A composite of the 8 anxiety items (a mean anxiety score) will be computed (1 [low anxiety score] - 5 [high anxiety score])
Change in perceived chronic pain social support from baseline to post-intervention to 1-month follow-up | Perceived chronic pain social support will be assessed at 3 timepoints: 1) baseline (i.e., at the start of the intervention), 2. post-intervention (i.e., immediately after the intervention), and 3. 1-month follow-up (30 days after the intervention ends)
  Diabetes Support Scale (Barrera, 2002), adapted for chronic pain: A summed score of the 12 support items will be computed (12-84, higher scores indicate greater support)
Change in anger from baseline to post-intervention to 1-month follow-up | Anger will be assessed at 3 timepoints: 1) baseline (i.e., at the start of the intervention), 2. post-intervention (i.e., immediately after the intervention), and 3. 1-month follow-up (30 days after the intervention ends)
  PROMIS Anger - Short Form 5a v1.1: A composite of the 5 anger items (a mean anger score) will be computed (1 [low anger score] - 5 [high anger score])
Change in self-efficacy for managing pain: PROMIS Self-Efficacy for Managing Symptoms v1.0 | Self-efficacy for managing pain will be assessed at 3 timepoints: 1) baseline (i.e., at the start of the intervention), 2. post-intervention (i.e., immediately after the intervention), and 3. 1-month follow-up (30 days after the intervention ends)
  PROMIS Self-Efficacy for Managing Symptoms v1.0 (10 items from the larger 30-item measure, adapted for self-efficacy for managing pain): A composite of the 10 self-efficacy items (a mean self-efficacy score) will be computed (1 [low self-efficacy score] - 5 [high self-efficacy score])
Change in helplessness | Helplessness will be assessed at 3 timepoints: 1) baseline (i.e., at the start of the intervention), 2. post-intervention (i.e., immediately after the intervention), and 3. 1-month follow-up (30 days after the intervention ends)
  Arthritis Helplessness Index (Nicassio et al., 1985), adapted for chronic pain: A summed score of the 15 helplessness items will be computed (15-60, higher scores indicate greater helplessness)
Change in self-efficacy for managing emotions: PROMIS Self-Efficacy for Managing Emotions - Short Form 4a v1.0 | Self-efficacy for managing emotions will be assessed at 3 timepoints: 1) baseline (i.e., at the start of the intervention), 2. post-intervention (i.e., immediately after the intervention), and 3. 1-month follow-up (30 days after the intervention ends)
  PROMIS Self-Efficacy for Managing Emotions - Short Form 4a v1.0: A composite of the 4 self-efficacy items (a mean self-efficacy score) will be computed (1 [low self-efficacy score] - 5 [high self-efficacy score])
Change in social isolation | Social isolation will be assessed at 3 timepoints: 1) baseline (i.e., at the start of the intervention), 2. post-intervention (i.e., immediately after the intervention), and 3. 1-month follow-up (30 days after the intervention ends)
  PROMIS - Social Isolation - Short Form 8a v2.0: A composite of the 8 social isolation items (a mean social isolation score) will be computed (1 [low social isolation score] - 5 [high social isolation score])
Change in pain catastrophizing: Pain Catastrophizing Scale | Pain catastrophizing will be assessed at 3 timepoints: 1) baseline (i.e., at the start of the intervention), 2. post-intervention (i.e., immediately after the intervention), and 3. 1-month follow-up (30 days after the intervention ends)
  Pain Catastrophizing Scale (Sullivan et al., 1995): A summed score of the 13 catastrophizing items will be computed (0-52, higher scores indicate greater catastrophizing)
Change in alexithymia | Alexithymia will be assessed at 3 timepoints: 1) baseline (i.e., at the start of the intervention), 2. post-intervention (i.e., immediately after the intervention), and 3. 1-month follow-up (30 days after the intervention ends)
  Toronto Alexithymia Scale (TAS-20): A summed score of the 20 alexithymia items will be computed (20-100, higher scores indicate greater alexithymia)
Change in substance use | Substance use will be assessed at 3 timepoints: 1) baseline (i.e., at the start of the intervention), 2. post-intervention (i.e., immediately after the intervention), and 3. 1-month follow-up (30 days after the intervention ends)
  Substance use questionnaire: 4 question-set recommended by the NIAAA (adapted for the "past week"): 1) Frequency of drinking / opioid use / marijuana use (0 [never] - 5 [every day]), 2) Number of drinks (0 [no drinks] - 10 [25 or more drinks]), 3) Maximum drinks (0 [no drinks] - 10 [36 or more drinks], 4) Frequency of binge drinking (0 [never] - 5 [every day])
Perceived emotional support within the Facebook group | Perceived emotional support within the Facebook group will be assessed at post-intervention (i.e., immediately after the intervention)
  PROMIS - Emotional Support - Short Form 8a, adapted for in-group support: A composite of the 8 emotional support items (a mean emotional support score) will be computed (1 [low emotional support score] - 5 [high emotional support score])

OTHER OUTCOMES:
Ambivalence over emotional expression | Ambivalence over emotional expression will be assessed at baseline (i.e., at the start of the intervention)
  Ambivalence Over Emotional Expressiveness Questionnaire (King & Emmons, 1990): A composite of the 14 ambivalence items (a mean ambivalence score) will be computed (1 [low ambivalence score] - 5 [high ambivalence score])
Perceived social constraints | Perceived social constraints will be assessed at baseline (i.e., at the start of the intervention)
  General Social Constraints Scale (Lepore & Ituarte, 1999): A summed score of the 15 social constraints items will be computed (15-60, higher scores indicate greater perceived social constraints)
Childhood adverse events | Childhood adverse events will be assessed at baseline (i.e., at the start of the intervention)
  Adverse Childhood Experience (ACE) Questionnaire: A summed score of the 10 ACE items will be computed (0-10, higher scores indicate greater adverse childhood experiences)
Attachment style | Attachment style will be assessed at baseline (i.e., at the start of the intervention)
  Experiences in Close Relationships Scale - Revised (ECR_R), avoidance items only (18 items): A composite of the 18 avoidance items (a mean avoidance score) will be computed (1 [low avoidance score] - 7 [high avoidance score])

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tankha H, Pester BD, Brumley KM, Cano A, Tong S, Grekin E, Bruinsma J, Gootee J, Lumley MA. A mixed-methods investigation into the us versus them mentality in Facebook groups for chronic pain. Health Psychol. 2023 Jul;42(7):460-471. doi: 10.1037/hea0001289. Epub 2023 May 4. PMID 37141005
- [Derived] Pester BD, Tankha H, Cano A, Tong S, Grekin E, Bruinsma J, Gootee J, Lumley MA. Facing Pain Together: A Randomized Controlled Trial of the Effects of Facebook Support Groups on Adults With Chronic Pain. J Pain. 2022 Dec;23(12):2121-2134. doi: 10.1016/j.jpain.2022.07.013. Epub 2022 Sep 9. PMID 36096353